CLINICAL TRIAL: NCT04322721
Title: Coagulopathy on the First Postoperative Day Predicts the Long-term Survival of Traumatic Brain Injury Patients: A Retrospective Cohort Study
Brief Title: Coagulopathy on the First Postoperative Day Predicts the Long-term Survival of Traumatic Brain Injury Patients
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDSJWKTBISC
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Traumatic Brain Injury; Coagulation Disorder
Keywords: Traumatic Brain Injury; Coagulation Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to identify the relationship between coagulopathy during the perioperative period (before the operation and on the first day after the operation) and the long-term survival of traumatic brain injury patients undergoing surgery, as well as to explore the predisposing risk factors that may cause perioperative coagulopathy.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is one of the leading causes of death and disability worldwide, and it represents a global health concern and financial burden [1, 2]. The main causes of early death in trauma victims are acidosis, hypothermia and coagulopathy, which are related to each other and influence each other. Thus, this vicious circle is often referred to as the " trauma triangle of death " [3, 4]. Trauma-induced coagulopathy manifests as a state of hypercoagulopathy trending towards thrombosis [5] and a state of hypocoagulopathy with progressive intracranial hemorrhage and increased systemic bleeding [6, 7].

There are many studies continuously proving that trauma-induced coagulopathy is common in traumatic brain injury patients [8-10] and the incidence of coagulation disorders has great heterogeneity, ranging from 7% to 54% [11, 12]. Reasons that cause this variation include the different techniques and definitions used, the heterogeneity of the patients and the various testing times [13]. Secondary coagulopathy after traumatic brain injury represent an important factor for unfavorable prognosis [14, 15], resulting in a nine-fold higher risk of death and a 30-fold higher risk of poor prognosis than in TBI patients without secondary coagulation disorder [7, 9, 16]. Mortality in TBI patients with coagulopathy is also highly heterogeneous, ranging from 22% to 66% [17, 18]. TBI patients with coagulopathy tend to suffer from delayed or progressive intracranial hemorrhage, as well as from microvascular thrombosis [19, 20].

Many retrospective and observational studies have focused on coagulation upon admission or the presence of any coagulation disorders during the whole period of hospitalization [21, 22]. A multicenter study described the course of coagulopathy in patients with isolated TBI, and associated it with CT characteristics and outcomes [15]. The previous study mostly focused on the coagulopathy on admission, while the association between coagulopathy in perioperative period and long-term survival of TBI patients has not been explored. It is important to explore this relationship because many TBI patients require surgical treatment, and it has been well established that the surgical intervention have an impact on the coagulation functions. We therefore investigated for the first time whether coagulopathy during the perioperative period, with the use of coagulation function tests performed before the operation and on the first day after the operation, was related to the long-term survival of these patients. Furthermore, we investigated the predisposing risk factors that may cause coagulopathy in the perioperative period, to the extent that these risk factors could be controlled and managed for avoiding coagulopathy.

ELIGIBILITY:
Inclusion Criteria:

1. The interval between injury and admission is less than 24 hours
2. Age>18yrs and age<80yrs
3. Non-head abbreviated injury score < 3
4. Did not undertake treatment before enrollment

Exclusion Criteria:

1. Take anticoagulants or antiplatelet drugs
2. Hemorrhagic or ischemic cerebrovascular disease occurred within six months
3. Other systemic diseases: uremia, cirrhosis, malignant tumor, etc

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The clinical data of TBI patients were retrospectively collected from January 1, 2015 to April 25, 2019 in the Second Affiliated Hospital of the Fourth Military Medical University. We included patients who recorded an intracranial injury as the main diagnosis or the coexisting diagnoses upon admission. Intracranial injuries were identified by WHO ICD-11 codes from NA07.0 to NA07.9.
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 3 month after onset
  The mortality rate of traumatic brain injury (TBI) patients undertook surgery at 3 month
Mortality | 12 month after onset
  The mortality rate of traumatic brain injury (TBI) patients undertook surgery at 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Dadhwal US, Pathak N. Damage Control Philosophy in Polytrauma. Med J Armed Forces India. 2010 Oct;66(4):347-9. doi: 10.1016/S0377-1237(10)80015-2. Epub 2011 Jul 21. PMID 27365740
- [Background] Mitra B, Tullio F, Cameron PA, Fitzgerald M. Trauma patients with the 'triad of death'. Emerg Med J. 2012 Aug;29(8):622-5. doi: 10.1136/emj.2011.113167. Epub 2011 Jul 23. PMID 21785151
- [Background] Chen H, Xue LX, Guo Y, Chen SW, Wang G, Cao HL, Chen J, Tian HL. The influence of hemocoagulation disorders on the development of posttraumatic cerebral infarction and outcome in patients with moderate or severe head trauma. Biomed Res Int. 2013;2013:685174. doi: 10.1155/2013/685174. Epub 2013 Aug 4. PMID 23984395
- [Background] Laroche M, Kutcher ME, Huang MC, Cohen MJ, Manley GT. Coagulopathy after traumatic brain injury. Neurosurgery. 2012 Jun;70(6):1334-45. doi: 10.1227/NEU.0b013e31824d179b. PMID 22307074
- [Background] Maegele M, Schochl H, Menovsky T, Marechal H, Marklund N, Buki A, Stanworth S. Coagulopathy and haemorrhagic progression in traumatic brain injury: advances in mechanisms, diagnosis, and management. Lancet Neurol. 2017 Aug;16(8):630-647. doi: 10.1016/S1474-4422(17)30197-7. Epub 2017 Jul 11. PMID 28721927
- [Background] Stein SC, Smith DH. Coagulopathy in traumatic brain injury. Neurocrit Care. 2004;1(4):479-88. doi: 10.1385/NCC:1:4:479. PMID 16174954
- [Background] Harhangi BS, Kompanje EJ, Leebeek FW, Maas AI. Coagulation disorders after traumatic brain injury. Acta Neurochir (Wien). 2008 Feb;150(2):165-75; discussion 175. doi: 10.1007/s00701-007-1475-8. Epub 2008 Jan 2. PMID 18166989
- [Background] Zhang J, Jiang R, Liu L, Watkins T, Zhang F, Dong JF. Traumatic brain injury-associated coagulopathy. J Neurotrauma. 2012 Nov 20;29(17):2597-605. doi: 10.1089/neu.2012.2348. Epub 2012 Oct 31. PMID 23020190
- [Background] Chhabra G, Rangarajan K, Subramanian A, Agrawal D, Sharma S, Mukhopadhayay AK. Hypofibrinogenemia in isolated traumatic brain injury in Indian patients. Neurol India. 2010 Sep-Oct;58(5):756-7. doi: 10.4103/0028-3886.72175. PMID 21045504
- [Background] Greuters S, van den Berg A, Franschman G, Viersen VA, Beishuizen A, Peerdeman SM, Boer C; ALARM-BLEEDING investigators. Acute and delayed mild coagulopathy are related to outcome in patients with isolated traumatic brain injury. Crit Care. 2011;15(1):R2. doi: 10.1186/cc9399. Epub 2011 Jan 5. PMID 21208418
- [Background] Kumar MA, Cao W, Pham HP, Raju D, Nawalinski K, Maloney-Wilensky E, Schuster J, Zheng XL. Relative Deficiency of Plasma A Disintegrin and Metalloprotease with Thrombospondin Type 1 Repeats 13 Activity and Elevation of Human Neutrophil Peptides in Patients with Traumatic Brain Injury. J Neurotrauma. 2019 Jan 15;36(2):222-229. doi: 10.1089/neu.2018.5696. Epub 2018 Aug 14. PMID 29848170